CLINICAL TRIAL: NCT04968899
Title: Intravenous Immunoglobulin Plus Oral Prednisone or High-dose Dexamethasone, for Adults With Immune Thrombocytopenia (ITP) With Moderate and Severe Bleeding: a Randomized, Multicentre Trial
Brief Title: IgIV Plus Prednisone vs High-dose Dexamethasone for ITP
Acronym: IVIORDEX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200017; 2021-000292-37 (EudraCT Number)
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Immune Thrombocytopenia (ITP)
Keywords: Immune thrombocytopenia (ITP); Dexamethasone; IntraVenous Immunoglobulin; Prednisone
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Dexamethasone; Immunoglobulins, Intravenous; Octagam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Oral dexamethasone (Neofordex®) 40 mg (Day1 to Day 4), ± an additional 4-days cycle of dexamethasone between days 10 and 21
  Interventions: Drug: Neofordex®
- Control (Active Comparator): IVIg (1g/kg D1-D2) plus prednisone (1 mg/kg/day x 21 days (3 weeks))
  Interventions: Drug: Intravenous immunoglobulins

INTERVENTIONS:
Drug: Neofordex® — Oral dexamethasone (Neofordex®) 40 mg (Day1 to Day 4), ± an additional 4-days cycle of dexamethasone between days 10 and 21.
  Other Names: Dexamethasone
  Arms: Experimental group
Drug: Intravenous immunoglobulins — IVIg (1g/kg D1-D2) plus oral prednisone (1 mg/kg/day x 21 days (3 weeks))
  Other Names: Tegeline®; Clayrig®,; Gammagard®,; Octagam®,; Privigen®,; Other IgIV patent medicine
  Arms: Control

SUMMARY:
ITP patients with low platelet count and active bleeding symptoms are at risk of life-threatening bleeding and therefore require a treatment with a rapid effect, reliable, and sustained. The combination of intravenous immunoglobulin (IVIg) and prednisone (1 mg/kg per day), is more rapidly and more frequently effective than high dose methylprednisolone to increase the platelet count. This combination is therefore usually given in patients with platelets count < 20 x 109/L and moderate to severe bleeding manifestations. Based on common practice in France and on French ITP guidelines, on average 50 % of patients with ITP and profound thrombocytopenia do actually receive IVIg (mostly during the initial phase of the disease) corresponding to approximately 1,500 ITP patients per year in France.

Whereas IVIg is usually well tolerated, renal insufficiency and congestive heart failure may occur, moreover IVIg are costly and non-easily available with supply difficulties in many countries including France.

High dose dexamethasone (DXM) (ie: 40 mg/d for 4 days) has recently emerged as a promising treatment for ITP. One recent meta-analysis as well as a controlled prospective trial suggest that the initial overall response was higher (> 80 %) and the time to response was shorter with dexamethasone (DXM) 40 mg/d given for 4 days compared to standard prednisone.

The investigators hypothesize that DXM could be a reasonable non-inferior alternative to IVIg, more convenient for patients with less adverse events and economically cost-effective for patients with moderate and severe bleeding manifestations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years ≤ 80 years
* Diagnosis of ITP whatever the duration of the disease (newly diagnosed or relapsed) according to the standard definition
* Platelet count ≤ 20 x 109/L
* Any cutaneous and/or any mucosal bleeding manifestations
* Affiliated to a social security regime
* Written consent from patient

Exclusion Criteria:

* Symptomatic COVID-19 disease
* Life-threatening bleeding defined as Intracranial hemorrhage and/or active organ bleeding (GI tract, urinary tract or menorrhagia with at least a 2 g/dl decrease of hemoglobin value from baseline).
* Ongoing anticoagulation treatment (Therapeutic Low molecular weight heparins (LMWHs), direct oral anticoagulants (DOACs) and vitamin K antagonists (VKAs))
* Previous non-response to IVIg or DEX
* Treatment with prednisone (1 mg/kg per day) for more than 3 days
* Any, contraindications to the prescribed Ig IV or prednisone patent medicine and to Neofordex®
* Ongoing severe infection
* Severe Renal insufficiency (DFG < 45 ml.min.1.73m2)
* Severe Cardiac insufficiency (FEVG < 30 %)
* Ongoing viral infection (uncontrolled HIV, Viral hepatitis, herpes, varicella, zona).
* Uncontrolled diabetes (Acido-cetosis)
* Psychotic state not yet controlled by treatment
* Inability or refusal to understand or refusal to sign the informed consent from study participation
* Persons deprived of their liberty by judicial or administrative decision,
* Persons under legal protection (guardianship, curatorship)
* Pregnant or breastfeeding woman or ineffective contraception
* Participation in another interventional study involving human participants or being in the exclusion period at the end of a previous study involving human participants.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2025-04-09 (Estimated); Study Completion 2026-10-09 (Estimated)

PRIMARY OUTCOMES:
Time to achieve an initial response (R) within 5 days. | 5 days

SECONDARY OUTCOMES:
Time to achieve an initial complete response (CR) in the two arms | between Day 1 and Day 5
  complete response (CR): defined by a platelet count > 100 x 109/L in the absence use of any other ITP directed therapies between Day 1 and Day 5
Duration of overall response from Day 1 to the end of the study in the two arms. | Day 1 to 6 months
Proportion of early treatment switches across arms | before day 5
Number of new bleeding manifestations between Day 1 and Day 5 in the two arms. | between Day 1 and Day 5
Rates of response (R) and complete response (CR) in the two arms. | at Day 28 and at 6 months
Number of new bleeding manifestations in the two arms. | Between Day 5 and Day 28
Number of adverse events in the two arms. | up to 6 months
Number of responders in patients with positive and negative anti-platelets antibodies in the two arms. | At 6 months
Number of outcome in patients with positive and negative anti-platelets antibodies in the two arms. | At 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION